CLINICAL TRIAL: NCT02281604
Title: In-line Filters on ICU
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Professor Kai Zacharowski, M.D., Ph.D., FRCA, Prof. Dr. Dr. med., Johann Wolfgang Goethe University Hospital
Other Study IDs: In-line Filter 13/14
Record Dates: First submitted 2014-10-29; First posted 2014-11-03 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Micropore Filters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 0.2/1.2 microliter filter: Use of 0.2/1.2 microliter filters for intravenous drug administration
- 5 mircroliter filter: Use of 5 microliter filters for intravenous drug administration

SUMMARY:
The purpose of this study is to determine whether the use of 0.2/1.2 microliter in-line filter reduces the incidence of severe vasoplegia comparing to the 5 microliter filter.

ELIGIBILITY:
Inclusion Criteria:

* all patients

Exclusion Criteria:

* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, which will be treated on the anaesthesiological/surgical ICU of the University Hospital Frankfurt between 2013 - 2014
Sampling Method: Non-Probability Sample
Enrollment: 3281 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Incidence of severe vasoplegia | participants will be followed for the duration of intensive care unit stay, an expected average of 1 week

SECONDARY OUTCOMES:
Organ dysfunction | participants will be followed for the duration of intensive care unit stay, an expected average of 1 week
  Severity of organdysfunction (SOFA-Score), incidence and severity of respiratory failure (Horovitz- Index), incidence and severity of acute kidney failure (RIFLE criteria), incidence and severity of delirium
Inflammation | participants will be followed for the duration of intensive care unit stay, an expected average of 1 week
  Interleukin-6
Duration of ICU and hospital stay | participants will be followed for the duration of intensive care unit/ hospital stay, an expected average of 1 or 4 week (s), respectively
In-hospital mortality | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Morbidity | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Incidence of preoperative myocardial infarction, stroke, pneumonia, sepsis and acute kidney failure according to routine documentation

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zacharowski, M.D., Principal Investigator — University Hospital Frankfurt. Department of Anesthesiology, Intensive-Care Medicine and Pain Therapy.

REFERENCES:
- [Derived] Schmitt E, Meybohm P, Herrmann E, Ammersbach K, Endres R, Lindau S, Helmer P, Zacharowski K, Neb H. In-line filtration of intravenous infusion may reduce organ dysfunction of adult critical patients. Crit Care. 2019 Nov 22;23(1):373. doi: 10.1186/s13054-019-2618-z. PMID 31757216